CLINICAL TRIAL: NCT05843773
Title: Low-Load Blood Flow Restriction Training With Patients Who Underwent a Total Knee Arthroplasty: a Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HES-SO Valais-Wallis (Other)
Collaborators: Leukerbad Clinic (Unknown); Berner Fachhochschule (BFH) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01102
Record Dates: First submitted 2023-03-07; First posted 2023-05-06 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-06

CONDITIONS: Total Knee Arthroplasty
Keywords: strength training; blood flow restriction; total knee arthroplasty

STUDY DESIGN:
Intervention Model Description: The present study is a feasibility study. The study is based on the Consort Checklist for pilot and feasibility trials. This will be a monocentric study; the patients will be recruited at the Leukerbad Clinic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Load Strength Training under Blood Flow Restriction (Experimental): Low Load Strength Training under blood flow restriction
  Interventions: Procedure: Low Load Strength Training under Blood Flow Restriction

INTERVENTIONS:
Procedure: Low Load Strength Training under Blood Flow Restriction — The first training includes one initiation/warm up set and two sets of normal training. Every set lasts 60 seconds and the patient is asked to bend and stretch the knee with a standard speed of 20°/s.
  From the second to the ninth training, the patient will have one warm up set plus three trainings sets. The speed of execution will be increased every training.
  The 20-40% range of the 1RM will be applied according to the values of the theoretical maximal strength.
  If no strength progression is observed in the three last training sessions, the speed of execution will automatically be increased by 15°/s.
  In order to keep the training intensity low and to not overload the knee, participants will be instructed to control the intensity with the Borg CR10. The volunteers will have to keep their efforts between 2/10 and 4/10. They will also be asked to stay in the range defined thanks to the theoretical maximal strength shown by the screen.

SUMMARY:
This project aims to investigate the feasibility of a low load (LL) isokinetic knee flexor and extensor strength training (ST) protocol under blood flow restriction (BFR) conditions in early postoperative total knee arthroplasty patients.

The intervention consists in testing an experimental strengthening protocol in the Leukerbad Clinic. 12 participants will be recruited and the intervention will last approximatively 3 weeks and will consist in 3 weekly ST.

The collected data will then be analysed and interpreted to define if such an intervention is feasible or not.

ELIGIBILITY:
Inclusion Criteria:

* Primary TKA surgery less than 12 days before inclusion
* Ability to participate fully in physiotherapy
* Ability to consent for study participation
* Age between 50 and 80 years old

Exclusion Criteria:

* Postoperative complication
* History of deep venous thrombosis
* History of vascular pathology
* History of metabolic condition
* Previous contralateral TKA
* Previous ipsilateral or contralateral total hip arthroplasty
* Any other lower extremity musculoskeletal chronic condition
* Any lower extremity injury within the last 6 months
* Pregnancy
* Sickle cell trait
* History of neurocognitive disorders
* Inability to follow the intervention protocol

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-01-06 (Actual)

PRIMARY OUTCOMES:
Practicality of the study protocol - Time to teach the protocol to the personnel | Before the beginning of the procedure
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: time needed to teach the protocol to the personnel in minutes
Practicality of the study protocol - Time needed for the pre-tests | Day 1 post-inclusion
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: time needed for the pre-tests in minutes
Practicality of the study protocol - Time needed for the post-tests | Day 1 post-inclusion
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: time needed for the post-tests in minutes; time needed for the intervention in minutes; human resources needed. We will also appraise the recruitment rates by evaluating the number of volunteers recruited within 6 months. We will then assess the retention rates by counting the number of dropouts and analysing the compliance/adherence rates. And finally, we will evaluate the costs by considering the equipment, recruitment, ethical commission, and human resources costs.
Practicality of the study protocol - Time needed for the post-tests | Last day of the intervention
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: time needed for the post-tests in minutes
Practicality of the study protocol - Time needed for the intervention | During the procedure (approximatively 3 weeks long)
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: time needed for the intervention in minutes
Practicality of the study protocol - Human ressources needed | During the procedure (approximatively 3 weeks long)
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: human resources needed.
Practicality of the study protocol - Recruitment rates | During the recruitment period (6months)
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: the recruitment rates by evaluating the number of volunteers recruited within 6 months.
Practicality of the study protocol - Retention rates | During the recruitment period (6months)
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: the retention rates by counting the number of dropouts and analysing the compliance/adherence rates. And finally, we will evaluate the costs by considering the equipment, recruitment, ethical commission, and human resources costs.
Practicality of the study protocol - Costs | From date of acceptation of the project (April 2022) to the anticipated end of the project (December 2023), assessed up to 90 weeks
  The term practicality refers to "the extent to which an intervention can be delivered when resources, time, commitment, or some combinations thereof are constrained in some way" (Bowen et al., 2009). We will therefore assess the ability of therapists to carry out the tests and intervention by evaluating the following variable: the costs by considering the equipment, recruitment, ethical commission, and human resources costs.
Acceptability of the intervention | Up to three weeks (duration of the intervention)
  The domain acceptability focuses on how the individuals involved in the study react to the intervention (Bowen et al., 2009). We will assess both the satisfaction with the intervention protocols and the perceived positive and negative effects during and after the intervention protocols. Both outcomes will be evaluated with the visual analogue scale (VAS).

SECONDARY OUTCOMES:
Preliminary data on benefits - Strength | During the procedure (approximatively 3 weeks long)
  The domain preliminary data on benefits refers to the effect of the intervention protocol that we will measure. For the outcome strength, we will measure the maximal strength of the knee flexors and extensors. The data assessed will be described in Newton meter (Nm) and will be gathered on the isokinetic dynamometer.
Preliminary data on benefits - Pain | During the procedure (approximatively 3 weeks long)
  The domain preliminary data on benefits refers to the effect of the intervention protocol that we will measure.
  The outcome pain will be measured with the Visual Analogue Scale. We will ask the patient before, between and after every set what is the rating and analyse it in the end of the study.
Preliminary data on benefits - Functionality | Up to three weeks (duration of the intervention)
  The domain preliminary data on benefits refers to the effect of the intervention protocol that we will measure.
  The outcome functionality will be assessed with the Knee Injury and Osteoarthritis Outcome Score (KOOS).
Preliminary data on benefits - Functionality | Up to three weeks (duration of the intervention)
  The domain preliminary data on benefits refers to the effect of the intervention protocol that we will measure.
  The second outcome for functionality will be assessed the 6 Minute Walk Test (6MWT).

CONTACTS AND LOCATIONS:
Locations (1):
- HES-SO, Sion, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No